CLINICAL TRIAL: NCT02761122
Title: Implication of Human Papillomavirus (HPV) in Lichen Physiopathology in Human
Brief Title: Implication of Human Papillomavirus (HPV) in Lichen Physiopathology in Human (HPVLichen)
Acronym: HPVLichen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: Société de Dermatologie Française (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-058; ID-RCB number : 2015-A01697-42 (Other: French national registration number of the study)
Record Dates: First submitted 2016-04-22; First posted 2016-05-04 (Estimated); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Lichen Planus
MeSH Terms: conditions — Lichen Planus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with lichen (Experimental): Patients with non-erosive lichen planus, erosive lichen planus or lichen sclerosus.
  Human biological samples :
  * Blood sample
  * Skin or mucosal brushing
  * Skin or mucosal biopsy
  Interventions: Procedure: Human biological samples

INTERVENTIONS:
Procedure: Human biological samples — * Blood sample
  * Skin or mucosal brushing
  * Skin or mucosal biopsy

SUMMARY:
Lichen planus is a chronic cutaneous and mucosal disease characterized by the infiltration of cluster of differentiation (CD) CD8 T lymphocytes, localized under the basal membrane and associated with apoptosis of basal keratinocytes, suggesting a reactivity of T lymphocytes toward keratinocyte antigen(s), so far unidentified. In a recent study, the research team at Institut Pasteur has demonstrated in a peculiar clinical form of lichen planus (erosive lichen planus), that the immunogenic target of CD8 T lymphocytes could be the immunodominant peptide of Human Papilloma Virus (HPV) 16.

In line with this recent work which shows for the first time a link between HPV-16 and an autoimmune disease, erosive lichen planus, the aim of te study is to test the hypothesis that HPV could be also involved in the pathogenesis of other clinical forms of lichen, such as non erosive lichen planus or lichen sclerosus.

DETAILED DESCRIPTION:
Lichen planus is a chronic cutaneous and mucosal disease characterized by the infiltration of cluster of differentiation (CD) CD8 T lymphocytes, localized under the basal membrane and associated with apoptosis of basal keratinocytes, suggesting a reactivity of T lymphocytes toward keratinocyte antigen(s), so far unidentified. In a recent study, the research team at Institut Pasteur has demonstrated in a peculiar clinical form of lichen planus (erosive lichen planus), that the immunogenic target of CD8 T lymphocytes could be the immunodominant peptide of Human Papilloma Virus (HPV) 16.

In line with this recent work which shows for the first time a link between HPV-16 and an autoimmune disease, erosive lichen planus, the aim of te study is to to test the hypothesis that HPV could be also involved in the pathogenesis of other clinical forms of lichen, such as non erosive lichen planus or lichen sclerosus.

Regarding erosive lichen planus, the aim is to test the cytotoxic function of the previously identified CD8 T lymphocytes specific for HPV16 E711-20.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 year-old
* Clinically or histologically confirmed lichen : Non-erosive lichen planus, Erosive lichen planus, or Sclerosus lichen
* At diagnosis of desease before treatment, or during flares of the disease, with or without intake or topical application of immunosuppressants
* Affiliated or beneficiary of a social security system
* Informed and written consent

Exclusion Criteria:

* Under 18 year-old,
* Legal protection measures,
* Inability to consent
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-05-17 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-04-16 (Actual)

PRIMARY OUTCOMES:
The use of the different segments of the Vbeta gene assessed by quantitative PCR, and the distribution of the different sizes of the complementarity determining regions (CDR) CDR3 by immunoscope. | 2 years
  In patients with a non-erosive type of lichen and with a lichen sclerosus et atrophicus, the hypothesis for oligoclonal bias in the T-cell receptor repertoire on peripheral and in situ CD4 and CD8 T lymphocytes will be tested realizing, on the 2 sorted subpopulations, a study of the use of the different segments of the Vbeta gene using quantitative Polymerase Chain Reaction (PCR) and a study of the distribution study of the different sizes of the CDR3 using immunoscope method.
  Depending on whether or not bias in the T-cell receptor repertoire exists, the study will be continued by looking for the same repertoire bias in situ, on injury site (skin or mucous, depending on the clinical type of lichen), and the research of clonal sequences (or clonotypes) from RNA of patients after cloning and complete sequencing. If clonotype T CD8 Vbeta3 are identified in these types of lichen, their specificity to HPV16 E711-20 wil be assessed by flow cytometry.

SECONDARY OUTCOMES:
The functionality and the cytotoxicity of CD8 Vbeta3 peripheric T lymphocytes assessed by flow cytometry. | 2 years
  In patients with erosive lichen planus, the functionality and the cytotoxicity of CD8 Vbeta3 peripheric T lymphocytes will be assessed showing their ability to recognize and destroy a target carrier of HPV16 E711-20 peptide by flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Lise Gougeon, Study Director — Institut Pasteur
Locations (3):
- France (3):
  - Service de Dermatologie du CHU de Besançon, Besançon
  - Service de Dermatologie de l'hôpital Saint Louis, Paris
  - Service de Dermatologie du CHU de Reims, Reims

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Viguier M, Perals C, Poirier B, Battistella M, Aubin F, Bachelez H, Pretet JL, Gheit T, Tommasino M, Touze A, Gougeon ML, Fazilleau N. Human papilloma virus-16-specific CD8+ T-cell expansions characterize different clinical forms of lichen planus and not lichen sclerosus et atrophicus. Exp Dermatol. 2023 Jun;32(6):859-868. doi: 10.1111/exd.14788. Epub 2023 Mar 15. PMID 36922453